CLINICAL TRIAL: NCT04718428
Title: Standardized Sonographic Analysis of Nails in Psoriatic Arthritis and Healthy Controls: Feasibility, Reliability, Discriminative Performance, and Demographic and Clinical Associations
Brief Title: Sonographic Analysis of Nails in Psoriatic Arthritis and Healthy Controls
Acronym: NUSGI
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2017.242
Record Dates: First submitted 2020-12-30; First posted 2021-01-22 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Psoriatic Arthritis; Psoriatic Nail
Keywords: nail ultrasonography; psoriatic arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- psoriatic arthritis: Patients with psoriatic arthritis who met the CASPAR criteria and were 18-70 years old were included. Participants with infection of the nails to be examined, loss of nails, trauma history of the nails, having the habit of nail biting, peripheral neuropathy, peripheral vascular disease, another rheumatological disease, systemic infection, and pregnancy were excluded.
  Interventions: Diagnostic Test: Nail Ultrasonography
- healthy controls: A gender- and age-matched healthy controls were included. They were recruited from the healthy relatives of the hospital staff. Participants with infection of the nails to be examined, loss of nails, trauma history of the nails, having the habit of nail biting, peripheral neuropathy, peripheral vascular disease, any rheumatological disease, systemic infection, and pregnancy were excluded.
  Interventions: Diagnostic Test: Nail Ultrasonography

INTERVENTIONS:
Diagnostic Test: Nail Ultrasonography — The MyLab 60 (Esaote Biomedica Genoa, Italy) device and linear probe were used. Nails were examined in B-mode grayscale and power Doppler.

SUMMARY:
This study aims to identify the nail ultrasonography (NUSG) properties in patients with psoriatic arthritis (PsA) and healthy controls by a participant-based evaluation; to assess feasibility, reliability, and discriminative performances; to explore final scorings; and to determine associations between the NUSG scores and participant characteristics, including demographics and disease-related factors.

DETAILED DESCRIPTION:
NUSG is a visualization method suitable for evaluating the subunits of the nail. The main purpose of this study is to identify NUSG properties in patients with PsA and healthy controls. The investigators recruited patients with PsA according to the CASPAR criteria and sex- and age-matched healthy controls into the study. NUSG parameters were examined by grayscale and power Doppler techniques for all of the fingernails and first toenails (12 nails); and five scorings including nail plate impairment score (NPIs), nail plate thickness score (NPTs), nail bed thickness score (NBTs), nail thickness score (NTs), and the Doppler activity score (DAs) were calculated. The investigators compared the PsA and control groups in terms of the NUSG scorings and also documented the discriminative performances (with receiver operating characteristic curve analysis) of the scorings. Then, the feasibility and reliability analysis of the NUSG scorings were performed. Finally, the association between the NUSG scores and participant characteristics, including sex, age, body weight, height, labor market participation, smoking, hemoglobin, disease duration, history of dactylitis, current enthesitis, radiographic sacroiliitis, C reactive protein, minimal disease activity, Disease Activity Index for Psoriatic Arthritis, Nail Psoriasis Severity Index, and Psoriasis Area Severity Index were explored.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Psoriatic arthritis
* Healthy controls without any musculoskeletal disease
* Must be at the age of 18-70 years

Exclusion Criteria:

* Infection of the nails to be examined
* Loss of nails to be examined
* Trauma history of the nails to be examined
* Having the habit of nail-biting
* Peripheral neuropathy
* Peripheral vascular disease
* Any rheumatological disease, except psoriatic arthritis
* Systemic infection
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients met the CASPAR criteria and healthy controls had no inflammatory or mechanical musculoskeletal disease. Participants in the age range of 18-70 were included.
  The control group was recruited from the healthy relatives of the hospital staff.
  The PsA group was recruited from Marmara University Physical Medicine and Rehabilitation/Rheumatology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-10-14 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
The nail plate impairment score | Baseline (T0)
  The sonographic normal nail plate term indicates a trilaminar band of the nail plate with two hyperechoic layers separated by a hypoechoic one. The "nail plate impairment score" means the number of nails with impaired trilaminar band (plate) among the 12 nails (all hand nails and toenails). The score ranges between 0-12, with 0 indicating no plate impairments (better) and 12 reflecting the maximal prevalence of impairment (worse).
The nail plate thickness score | Baseline (T0)
  The plate thickness of each nail was measured (in millimeters) by greyscale USG, then, the sum of 12 nails evaluated (all hand nails and toenails) was calculated as "nail plate thickness score" for a participant (in millimeters). Higher scores were expected to mean worse outcome.
The nail bed thickness score | Baseline (T0)
  The sonographic nail bed is the dark area below the nail plate to the cortical bone. The nail bed thickness of each nail was measured (in millimeters) by greyscale USG, then, the sum of 12 nails evaluated (all hand nails and toenails) was calculated as "nail bed thickness score" (in millimeters) for a participant. Higher scores were expected to mean worse outcome.
The nail thickness score | Baseline (T0)
  The total nail thickness (including the plate and bed) of each nail was measured (in millimeters) by greyscale USG, then, the sum of 12 nails evaluated (all hand nails and toenails) was calculated as "nail thickness score" (in millimeters) for a participant. Higher scores were expected to mean worse outcome.
The Doppler activity score | Baseline (T0)
  Doppler activity of the nail bed and matrix was measured by power Doppler USG. The power Doppler signal for each nail was graded from 0 to 3: 1 point for a signal in less than 25 percent of the nail bed area, 2 points for a signal 25 to 50 percent, 3 points for a confluent signal in more than 50 percent of the nail bed area, and 0 point for no signal. Then, the sum of 12 nails evaluated (all hand nails and toenails) was calculated as "Doppler activity score". The score ranges between 0-36, with 0 indicating no activity (better) and 36 reflecting the maximal activity (worse).

SECONDARY OUTCOMES:
Interobserver reliability of the NUSG scorings | Baseline (T0)
  Patients with PsA were evaluated twice in order to assess interobserver reliability. For this purpose, another investigator experienced in musculoskeletal USG performed the ultrasonographic evaluations with the same device but separately from the one who made the first assessment. Then, the consistency between the observers was calculated for each scoring by intraclass correlation coefficient (range 0-1).
Intraobserver reliability of the NUSG scorings | Two weeks after the baseline (T1)
  Patients with PsA were evaluated again in order to assess intraobserver reliability. For this purpose, the same rheumatologist experienced in musculoskeletal USG performed the ultrasonographic evaluations again, after 2 weeks. Then, the consistency between the observers was calculated for each scoring by intraclass correlation coefficient (range 0-1).

OTHER OUTCOMES:
Minimal Disease Activity | Baseline (T0)
  "Minimal Disease Activity" is used for remission criteria in patients with PsA. It is defined as 5 out of 7 of the following criteria: tender joint count ≤1, swollen joint count ≤1, PASI ≤1, patient pain visual analog score (VAS) ≤15 mm, patient global disease activity VAS ≤20 mm, health assessment questionnaire ≤0.5, and tender entheseal points ≤1
Disease Activity index for PSoriatic Arthritis | Baseline (T0)
  "Disease Activity index for Psoriatic Arthritis" is used for disease activity states and response criteria in patients with PsA. It is simply calculated by summing swollen + tender joint counts + VAS pain + VAS patient global assessments + C reactive protein.
Psoriasis Area and Severity Index | Baseline (T0)
  "Psoriasis Area and Severity Index" is used for the measurement of severity of psoriasis. It combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease). The body is divided into four sections: head 10 percent, arms 20 percent, trunk 30 percent, legs 40 percent. Each of these areas is scored by itself, and then the four scores are combined into the final score. For each section, the percent of area of skin involved, is estimated and then transformed into a grade from 0 to 6 (0: 0 percent of involved area, 1: < 10 percent of involved area, 2: 10-29 percent of involved area, 3: 30-49 percent of involved area, 4: 50-69 percent of involved area, 5: 70-89 percent of involved area, 6: 90-100 percent of involved area) Within each area, the severity is estimated by three clinical signs: erythema, induration and desquamation.
Nail Psoriasis Severity Index | Baseline (T0)
  "Nail Psoriasis Severity Index" is used to measure the severity of inspectional nail psoriasis by area of involvement in the nail unit: Each nail is divided into four quadrants and any nail plate or bed changes found are accounted for, generating a score that varies from 1-80. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Tuncay Duruöz, Professor, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sandre MK, Rohekar S. Psoriatic arthritis and nail changes: exploring the relationship. Semin Arthritis Rheum. 2014 Oct;44(2):162-9. doi: 10.1016/j.semarthrit.2014.05.002. Epub 2014 May 6. PMID 24932889
- [Background] Arbault A, Devilliers H, Laroche D, Cayot A, Vabres P, Maillefert JF, Ornetti P. Reliability, validity and feasibility of nail ultrasonography in psoriatic arthritis. Joint Bone Spine. 2016 Oct;83(5):539-44. doi: 10.1016/j.jbspin.2015.11.004. Epub 2015 Dec 10. PMID 26688297
- [Derived] Acer Kasman S, Gezer HH, Baklacioglu HS, Erdem Gursoy D, Duruoz MT. A standardized sonographic analysis of nails in psoriatic arthritis and healthy controls: Feasibility, reliability, diagnostic performance, and demographic and clinical associations. Joint Bone Spine. 2021 Oct;88(5):105197. doi: 10.1016/j.jbspin.2021.105197. Epub 2021 Apr 24. PMID 33901660